CLINICAL TRIAL: NCT05321264
Title: Nursing Intervention in Adults to Promote Dengue Prevention and Control Behaviors
Brief Title: Educational Intervention to Promote Control Behaviors and Prevention of Dengue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-29
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-06

CONDITIONS: Dengue
Keywords: Standardized Nursing Terminology; Prevention & control; Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention is defined as educational support (improving the knowledge of the disease, identification of risks and consequences), behavioral support (promoting skills related to personal, home, and environmental self-care) and attitudinal support (reflecting on benefits and risks).
  Interventions: Behavioral: Educational nursing intervention
- Control (No Intervention): Control group will receive the usual strategy of a health service provider institution.

INTERVENTIONS:
Behavioral: Educational nursing intervention — Four weekly individualized intervention sessions, with a duration of 40 minutes.
  Arms: Intervention

SUMMARY:
This study will assess the effect of an educational nursing intervention in adults to promote dengue control and prevention behaviors, in comparison with the usual strategy of a health service provider institution. The intervention uses the Nola Pender Health Promotion Model as a theoretical framework. Findings will be assessed using the nursing outcomes "risk control" and "participation in health care decisions" from the Nursing Outcomes Classification (NOC).

DETAILED DESCRIPTION:
Annually, there are 390 million cases of dengue, mostly due to the inadequate application of sanitary behaviors in the management and control of the vector, having as background the lack of knowledge of the population in the appropriation and incorporation of sanitary measures in the different environments. In addition to the cognitive and behavioral component, dengue has cultural, political, social and economic causes.

The evidence indicates that, from health education, educational interventions have been developed to reduce the disease, but most of them have not been carried out in rural areas following a theoretical framework that guides the intervention that leads to an impact on health promoting behaviors.

The use of the NOC results makes it possible to visualize the impact of nursing care and constitute scientific support for the advancement of the nursing discipline.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old.
* Inhabitant of the rural area.
* Participant in health promotion and disease prevention programs.
* Initial score less than or equal to 3.5 on the NOC outcomes: risk control and participation in health care decisions.

Exclusion Criteria:

* People with a score less than or equal to 24 on the cognitive mini mental test.
* Incomplete registration of information in databases of a health service provider institution.
* People with dengue (dengue with warning signs, and severe dengue).
* People who do not have mobile phone availability.
* Illiterate people.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Risk control | 2 months
  NOC outcome. Personal actions to understand, prevent, eliminate, or reduce modifiable health threats. It includes indicators such as identifies risk factors, acknowledges ability to change behavior, develops effective risk control strategies, commits to risk control strategies and modifies lifestyle to reduce risk. This outcome will be evaluated by a Likert scale, being 1 the worst score and 5 best score.

SECONDARY OUTCOMES:
Participation in health care decisions | 2 months
  NOC outcome. Personal involvement in selecting and evaluating health care options to achieve desired outcome. It includes indicators such as identifies health outcome priorities, specifies health outcome preference and identifies barriers to desired outcome achievement. This outcome will be evaluated by a Likert scale, being 1 the worst score and 5 best score.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Canon Montanez, PhD, Study Director — Universidad de Antioquia
Locations (1):
- Yolima Judith Llorente Perez, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Llorente Perez YJ, Rodriguez-Acelas AL, Mattiello R, Canon-Montanez W. Effectiveness of a Nursing Educational Intervention in Adults to Promote Control Behaviors Against Dengue: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 23;13:e54286. doi: 10.2196/54286. PMID 38393755